CLINICAL TRIAL: NCT02396290
Title: Clinical Study on Efficacy and Safety of Platelet Rich Plasma Combined With Laser for Scar Treatment
Brief Title: Clinical Effect of Platelet Rich Plasma Combined With Laser on Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0998
Record Dates: First submitted 2015-03-09; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-07

CONDITIONS: Acne Scar
Keywords: acne scar; fractional carbon dioxide laser; platelet rich plasma
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fractional CO2 laser with PRP (Experimental): fractional carbon dioxide laser followed by intradermal injection of platelet rich plasma
  Interventions: Procedure: fractional carbon dioxide laser with platelet rich plasma
- fractional CO2 laser with NS (Active Comparator): fractional carbon dioxide laser followed by intradermal injection of NS
  Interventions: Procedure: fractional carbon dioxide laser with NS

INTERVENTIONS:
Procedure: fractional carbon dioxide laser with platelet rich plasma — fractional carbon dioxide laser followed by platelet rich plasma injection
  Other Names: COFRAX with autologous PRP
  Arms: fractional CO2 laser with PRP
Procedure: fractional carbon dioxide laser with NS — fractional carbon dioxide laser followed by normal saline injection
  Other Names: COFRAX with normal saline
  Arms: fractional CO2 laser with NS

SUMMARY:
Investigation of Clinical Effect of Platelet Rich Plasma Combined With Laser on Acne Scar

DETAILED DESCRIPTION:
Platelet Rich Plasma may relieve the adverse effect of laser treatment. and it can be expected to improve acne treatment result.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe acne scar

Exclusion Criteria:

* taken procedures for acne scar within 6 months
* underlying diabetes mellitus, keloid, or malignancy

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Global assessment of acne scar | 12 weeks
  5-point grading of acne scar

SECONDARY OUTCOMES:
ECCA (échelle d'évaluation clinique des cicatrices d'acné) | 12 weeks
  quantitative analysis of acne scar
adverse effect assessment | 12 weeks
  adverse effect assessment - erythema index, Epithelization Scale (0-12 point)

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, PhD, Study Chair — Department of Dermatology, Seoul National University College of Medicine; Seonguk Min, Msc, Principal Investigator — Department of Dermatology, Seoul National University College of Medicine
Locations (1):
- Department of Dermatology, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Tierney EP, Eisen RF, Hanke CW. Fractionated CO2 laser skin rejuvenation. Dermatol Ther. 2011 Jan-Feb;24(1):41-53. doi: 10.1111/j.1529-8019.2010.01377.x. PMID 21276157